CLINICAL TRIAL: NCT04519489
Title: The Efficacy of PAP Therapy on Reducing AF Recurrence in Patients With Morbidity of OSA: a Clinical Randomized Control Trial
Brief Title: The Efficacy of PAP Therapy on Reducing AF Recurrence in Patients With Morbidity of OSA
Acronym: AFOSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and investigators aligned to terminate this study.
Sponsor: Philips (China) Investment CO., LTD (Industry)
Collaborators: Peking University First Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); Beijing Tongren Hospital (Other); Fu Wai Hospital, Beijing, China (Other); Shanghai 6th People's Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICBE-2-29320
Record Dates: First submitted 2020-07-06; First posted 2020-08-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea
Keywords: Recurrence; Positive Airway Pressure
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PAP therapy with telemonitoring (Experimental): This arm will consist of 86 subjects.
  Interventions: Device: PAP therapy with telemonitoring
- Control group (Other): This arm will consist of 43 subjects.
  Interventions: Other: AF standard management and OSA general care

INTERVENTIONS:
Device: PAP therapy with telemonitoring — This study intends to investigate effect of PAP therapy on reducing AF recurrence rate in the patients in co-morbidity of OSA. The study will use 2 investigational devices: Philips DreamStation and Philips EncoreAnywhere. Philips DreamStation is used as the PAP therapy device to provide PAP therapy on the study subjects; Philips EncoreAnywhere is used as a telemonitoring service to provide monitoring by physicians that ensure good adherence to PAP. In addition, subjects in the intervention group will also receive AFib standard management and OSA general care.
  Arms: PAP therapy with telemonitoring
Other: AF standard management and OSA general care — Subjects in the control group will receive AF standard management and OSA general care. The treatment, medical care, and AF management for the subjects will be performed at the study hospitals following the newly updated Chinese AF management guideline 'Current knowledge and management recommendations of atrial fibrillation: 2018'.All subjects including the intervention group and the control group will receive the education materials to understand the disease, risk, and management of OSA. All subjects will also receive the general intervention for OSA, including suggestions for body weight control, smoking cessation, alcohol limiting, lateral position sleep, etc.
  Arms: Control group

SUMMARY:
This study aims to test the effectiveness of positive airway pressure therapy on reducing clinical failure after rhythm control treatment and restoring with regular heart beat in atrial fibrillation patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
This study aims to test the effectiveness of positive airway pressure therapy on reducing clinical failure after rhythm control treatment and restoring with regular heart beat in atrial fibrillation patients with obstructive sleep apnea. The study is designed as a multi-center randomized control trial, which plans to recruit 129 atrial fibrillation patients with obstructive sleep apnea (86 in the intervention group with atrial fibrillation standard care and positive airway pressure therapy, 43 in the control group with atrial fibrillation standard care but no positive airway pressure therapy). The subjects will in total visit the hospital 4 times during their 6 months follow-up period, at baseline, 1st, 3rd, and 6th month. Subjects will undergo questionnaire surveys and medical examinations at each visit. The primary objective is to compare after 6months, the clinical failure rate between the group with positive airway pressure therapy and the group with no positive airway pressure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent atrial fibrillation:

  1. Paroxysmal: at least having one episode every month for the last recent 6 months. Each episode with symptoms lasting for over 30 minutes and at least one episode is documented (≥30 seconds episode length, documented by ECG).
  2. Persistent: lasting over 7 days to 1 year persistent AF with ECG documented.
* Implement a rhythm control strategy, including:

  1. Ablation and restored on sinus rhythm after the procedure.
  2. Underwent medical or electrical cardioversion during hospitalization and restored on sinus rhythm before enrollment.
* OSA diagnosed with PSG test showing AHI≥10;
* 18 ≤ Age ≤ 75;
* Willing to participate in the study;
* Able to provide informed consent;
* Having access to smartphones and the internet, and be capable of using them.

Exclusion Criteria:

* BMI > 30 kg/m2;
* LVEF ≤ 40% or HF with NYHA III/ IV;
* Other atrial arrhythmias, atrial flatter;
* Myocardial infarction;
* Hypertrophic Cardiomyopathy (HCM);
* Congenital heart disease;
* A clear diagnosis with heart valve diseases (including moderate-severe mitral stenosis/ insufficiency, moderate-severe aortic stenosis/ insufficiency);
* Hyperthyroidism heart disease;
* Other acute diseases leading to temporary AF;
* In surgery perioperative period;
* Accepted other cardiothoracic surgery except for ablation;
* PSG test showing mainly central apneas (Cheyne-Stokes breathing);
* Pulmonary diseases causing dyspnea at rest or on minimal exertion;
* With other active major organ system disease that is not suitable for study participation, such as cancer, severe liver diseases, severe kidney diseases, etc.;
* With significantly impaired cognitive function, having severe problems in learning, memory, perception, and problem solving, and are unable to understand or not be competent to the informed consent;
* Having already accepted treatment to the sleep apnea syndrome;
* Having received intervention in any other trial within 30 days prior to the planned recruitment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with documented AFib recurrence | From baseline to the event occurs, up to 6 months.
  The primary outcome is number of participants with documented clinical failure. The documented clinical failure is defined as fulfilling any one of the following situations: documented recurrence of atrial fibrillation, atrial flutter or atrial tachycardia (lasting more than 30 seconds), new prescription of antiarrhythmic drugs (class I or III), repeat ablation (for patients underwent ablation at baseline) or new ablation (for patients used antiarrhythmic drugs for rhythm control at baseline).

SECONDARY OUTCOMES:
Change from baseline in atrial fibrillation burden at 6 months | Baseline, the 6th month.
  Atrial fibrillation burden from baseline to 6 months will be tested by single-lead ECG, calculated by total time in AF divided by the total time in sinus rhythm
Changes from baseline in self-rated AF symptoms at 1 month, 3 months and 6 months. | Baseline, the 1st month, 3rd month and 6th month.
  Self-rated AF symptoms will be tested with the modified EHRA Symptom Scale
Changes from baseline in quality of life at 3 months and 6 months. | Baseline, the 3rd month and 6th month.
  Quality of life will be tested with EQ-5D questionnaire
Changes from baseline in daytime sleepiness at 1 month, 3 months and 6 months. | The 1st month, 3rd month and 6th month.
  Sleepiness will be tested with the Epworth Sleepiness Scale (ESS).
Other cardiovascular events | From baseline to the event occurs, up to 6 months.
  Other cardiovascular events will be diagnosed and recorded by physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Ye, Professor, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Yong Huo, Professor, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaranov DM, Smyrlis A, Usatii N, Butler A, Petrini JR, Mendez J, Warshofsky MK. Effect of obstructive sleep apnea on frequency of stroke in patients with atrial fibrillation. Am J Cardiol. 2015 Feb 15;115(4):461-5. doi: 10.1016/j.amjcard.2014.11.027. Epub 2014 Nov 29. PMID 25529543
- [Background] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Li L, Wang ZW, Li J, Ge X, Guo LZ, Wang Y, Guo WH, Jiang CX, Ma CS. Efficacy of catheter ablation of atrial fibrillation in patients with obstructive sleep apnoea with and without continuous positive airway pressure treatment: a meta-analysis of observational studies. Europace. 2014 Sep;16(9):1309-14. doi: 10.1093/europace/euu066. Epub 2014 Apr 2. PMID 24696222
- [Background] Shukla A, Aizer A, Holmes D, Fowler S, Park DS, Bernstein S, Bernstein N, Chinitz L. Effect of Obstructive Sleep Apnea Treatment on Atrial Fibrillation Recurrence: A Meta-Analysis. JACC Clin Electrophysiol. 2015 Mar-Apr;1(1-2):41-51. doi: 10.1016/j.jacep.2015.02.014. Epub 2015 Apr 20. PMID 29759338
- [Background] Qureshi WT, Nasir UB, Alqalyoobi S, O'Neal WT, Mawri S, Sabbagh S, Soliman EZ, Al-Mallah MH. Meta-Analysis of Continuous Positive Airway Pressure as a Therapy of Atrial Fibrillation in Obstructive Sleep Apnea. Am J Cardiol. 2015 Dec 1;116(11):1767-73. doi: 10.1016/j.amjcard.2015.08.046. Epub 2015 Sep 12. PMID 26482182
- [Background] Nalliah CJ, Sanders P, Kalman JM. Obstructive Sleep Apnea Treatment and Atrial Fibrillation: A Need for Definitive Evidence. J Cardiovasc Electrophysiol. 2016 Aug;27(8):1001-10. doi: 10.1111/jce.12981. Epub 2016 May 31. PMID 27060686
- [Background] Craig S, Pepperell JC, Kohler M, Crosthwaite N, Davies RJ, Stradling JR. Continuous positive airway pressure treatment for obstructive sleep apnoea reduces resting heart rate but does not affect dysrhythmias: a randomised controlled trial. J Sleep Res. 2009 Sep;18(3):329-36. doi: 10.1111/j.1365-2869.2008.00726.x. Epub 2009 Jun 22. PMID 19549077
- [Background] Copur AS, Erik Everhart D, Zhang C, Chen Z, Shekhani H, Mathevosian S, Loveless J, Watson E, Kadri I, Wallace L, Simon E, Fulambarker AM. Effect of personality traits on adherence with positive airway pressure therapy in obstructive sleep apnea patients. Sleep Breath. 2018 May;22(2):369-376. doi: 10.1007/s11325-017-1559-5. Epub 2017 Aug 30. PMID 28856525
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Hurst NP, Kind P, Ruta D, Hunter M, Stubbings A. Measuring health-related quality of life in rheumatoid arthritis: validity, responsiveness and reliability of EuroQol (EQ-5D). Br J Rheumatol. 1997 May;36(5):551-9. doi: 10.1093/rheumatology/36.5.551. PMID 9189057
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Kilicaslan F, Verma A, Saad E, Themistoclakis S, Bonso A, Raviele A, Bozbas H, Andrews MW, Beheiry S, Hao S, Cummings JE, Marrouche NF, Lakkireddy D, Wazni O, Yamaji H, Saenz LC, Saliba W, Schweikert RA, Natale A. Efficacy of catheter ablation of atrial fibrillation in patients with hypertrophic obstructive cardiomyopathy. Heart Rhythm. 2006 Mar;3(3):275-80. doi: 10.1016/j.hrthm.2005.11.013. PMID 16500298
- [Background] Becker PH, Sperveslage H. Organochlorines and heavy metals in herring gull (Larus argentatus) eggs and chicks from the same clutch. Bull Environ Contam Toxicol. 1989 May;42(5):721-7. doi: 10.1007/BF01700394. No abstract available. PMID 2743002